CLINICAL TRIAL: NCT01021709
Title: Trial of Transcranial Direct Current Stimulation (tDCS) Using Alternative Electrode Montages
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09343
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Major Depression
Keywords: depression; direct current stimulation; extracephalic electrode
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tDCS with alternative electrode montage (Experimental): Treating major depression with either alternative tDCS electrode montage.
  Interventions: Device: tDCS (Eldith DC-Stimulator (CE certified))

INTERVENTIONS:
Device: tDCS (Eldith DC-Stimulator (CE certified)) — tDCS session lasting continuously for 20 minutes at 2 mA. Conductive rubber electrodes (7 x 5 cm = 35 cm2 & 10 x 10 cm = 100 cm2) covered by sponges soaked in saline will be used, held in place by a band. The current will be gradually increased to the level of 2 mA over 30 seconds (to avoid the sensation of a flash).
  Other Names: Eldith DC-Stimulator (CE certified)

SUMMARY:
Among antidepressant treatments, ECT stands as the most effective in treating acute depression. However, patient concerns with the cognitive side effects of ECT have encouraged the development of new and more focal forms of brain stimulation such as transcranial Direct Current Stimulation (tDCS). Our current study of tDCS as a treatment for depression suggests that this technique has antidepressant effects and is safe, painless and well tolerated. However, not all patients may respond to this treatment in the way that it is currently administered and the concern of possible relapse in some patients who respond to tDCS has raised interest in finding alternative, possibly more optimal ways of administering tDCS. This study will investigate whether using alternative electrode montages can improve the antidepressant effects of tDCS in people suffering from depression.

ELIGIBILITY:
Inclusion Criteria:

1. Subject met inclusion criteria for study HREC 07305 (a sham controlled study of transcranial direct current stimulation (tDCS) as a treatment for depression).
2. Subject completed study HREC 07305.
3. Subject either did not reach remission at the end of trial (defined as MADRS score of ≤ 10) or suffered an early relapse (within a month of finishing the trial).

Exclusion Criteria:

1. Diagnosis (as defined by DSM-IV) of: any psychotic disorder (lifetime); bipolar disorder; eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder current or within the past year); mental retardation.
2. History of drug or alcohol abuse or dependence (as per DSM-IV criteria) within the last 3 months (except nicotine and caffeine).
3. Inadequate response to ECT in the current episode of depression.
4. Subject is on regular benzodiazepine medication which it is not clinically appropriate to discontinue.
5. Subject requires a rapid clinical response due to inanition, psychosis or high suicide risk.
6. Neurological disorder or insult, e.g., recent stroke (CVA), which places subject at risk of seizure or neuronal damage with tDCS.
7. Subject has metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
8. Female subject who is pregnant, or of child-bearing age, sexually active and not using reliable contraception (urine test for pregnancy will be used).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS). | 6 months
  Baseline (pre-treatment), post 8, post 15 and post 20 tDCS sessions, and follow-up 1 week, 1 month, 3 months and 6 months post treatment

SECONDARY OUTCOMES:
Inventory of Depressive Symptomatology (IDS-C). | 6 months
  Baseline (pre-treatment), post 8, post 15 and post 20 tDCS sessions, and follow-up 1 week, 1 month, 3 months and 6 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute, University of New South Wales, Sydney, New South Wales, Australia

REFERENCES:
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au